CLINICAL TRIAL: NCT02272127
Title: Intercalated Combination of Chemotherapy Plus Icotinib for Patients Undergoing Resection of EGRF Mutation-positive Non-small-cell Lung Cancer
Brief Title: Study of Chemotherapy Plus Icotinib to Treat EGFR Mutation-positive Non-small-cell Lung Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Principal Investigator, Kaican Cai, Chief Physician，Associate Professor, Nanfang Hospital, Southern Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NFEC-2014-069
Record Dates: First submitted 2014-09-27; First posted 2014-10-22 (Estimated); Last update posted 2014-10-22 (Estimated); Status verified 2014-10

CONDITIONS: NSCLC
Keywords: EGFR tyrosine kinase inhibitor
MeSH Terms: interventions — icotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- intercalated treatment (Experimental): Patients will receive 4 cycles treatment: chemotherapy(day 1) plus intercalated icotinib(day 8-21) every 3 weeks, and then oral icotinib continuously for 2 years or until disease progression or unacceptable toxic effects
  Interventions: Drug: icotinib

INTERVENTIONS:
Drug: icotinib

SUMMARY:
Non-small-cell lung cancer (NSCLC) patients with activating epidermal growth factor receptor (EGFR) mutations are exquisitely sensitive to epidermal growth factor receptor tyrosine kinase inhibitors (EGFR-TKIs) which is widely used in advanced patients. Whether treatment with EGFR-TKIs improves outcomes in patients with resected NSCLC harboring EGFR mutations is still under investigated. This study aims to observe and compare the efficacy and safety of intercalated combination of chemotherapy plus icotinib in patients undergoing resection of EGRF mutation-positive non-small cell lung cancer stagingⅠB (with high risk factor) to ⅢA.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing completely resection of EGRF mutation-positive NSCLC
* Staging ⅠB (with high risk factor) to ⅢA
* PS<2
* Adequate hematological, biochemical and organ functions.

Exclusion Criteria:

* Systemic anticancer therapy prior to surgery, other malignancies before or during the study, any unstable illness, women who were pregnant or lactating.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2014-07; Primary Completion 2017-07 (Estimated); Study Completion 2019-07 (Estimated)

PRIMARY OUTCOMES:
Disease free survival | from the date of surgery until the date of first confirmed disease relapse or metastasis, assessed up to 5 years

SECONDARY OUTCOMES:
Number of Participants with Adverse Effects | duration of receiving chemotherapy and oral icotinib, expected to be 2.5 years

CONTACTS AND LOCATIONS:
Overall Officials: Kaican Cai, MD, Principal Investigator — Nanfang Hospital, Southern Medical University
Locations (1):
- Nanfang Hospital of Southern Medical University, Guangzhou, Guangdong, China